CLINICAL TRIAL: NCT00758134
Title: Prospective Phase II Trial Evaluating Efficacy of Trastuzumab Therapy in HER2 FISH Positive and/or HER2 Mutation Positive, Pretreated, Non-Small Cell Lung Cancer Patients (MO20509)
Brief Title: Trastuzumab Therapy in Non-Small Cell Lung Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, MD, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2007-001; 2007-003709-29
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: NON-SMALL CELL LUNG CANCER
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Trastuzumab 6 mg/Kg
  Interventions: Drug: Trastuzumab (Herceptin)

INTERVENTIONS:
Drug: Trastuzumab (Herceptin) — Trastuzumab 6 mg/Kg every 3 weeks i.v. (loading dose 8 mg/Kg i.v.)
  Other Names: Herceptin

SUMMARY:
This is a prospective study assessing efficacy of trastuzumab therapy in pretreated NSCLC patients. Patients with locally advanced or metastatic NSCLC, HER2 FISH positive and/or with HER2 gene mutation, pretreated with at least one previous chemotherapy line will be considered eligible for the trial. After evaluation of inclusion and exclusion criteria, and after signature of informed consensus form, all eligible patients will receive trastuzumab 6 mg/kg every 3 weeks (8 mg/kg loading dose) until disease progression, unacceptable toxicity or patient refusal.

ELIGIBILITY:
Inclusion Criteria:

* • Histologically confirmed diagnosis of NSCLC. Availability of tumor tissue for HER2 FISH analysis and/or HER2 gene mutation analysis is mandatory

  * Stage IIIB (with effusion) or stage IV or disease relapsed after surgery or radiotherapy and in any case not suitable for radiotherapy or surgery with curative intent
  * HER2 FISH positive defined as high polysomy or gene amplification, or presence of HER2 gene mutation in exon 20
  * At least one measurable lesion
  * Patients pretreated with at least one chemotherapy regimen. Previous therapy with erlotinib or other tyrosine kinase inhibitors is allowed.
  * Patients compliance to trial procedures
  * Age ≥ 18 years
  * Written informed consent
  * Adequate BM function (ANC ≥1.5x109/L, Platelets ≥100x109/L, HgB >9 g/dl)
  * Adequate liver function (bilirubin <G2, transaminases no more than 3xULN/<5xULN in present of liver metastases).
  * Normal level of alkaline phosphatase and creatinine
  * If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of approved contraceptive method [intrauterine contraceptive device (IUD), birth control pills, or barrier device] during and for three months after trial.
  * ECOG performance status 0-1 and life expectancy of at least 3 months
  * Have recovered from the acute, reversible effects of prior surgery or radiotherapy. This means that at least 3 weeks should have elapsed since prior radiotherapy.

Exclusion Criteria:

* • HER2 FISH negative tumor and no evidence of HER2 gene mutation in exon 20

  * Concomitant radiotherapy
  * Untreated brain metastases or leptomeningeal disease involvement.
  * All disease sites previously included in radiotherapy fields. If all sites were included in radiotherapy fields patient is eligible only if there is evidence of progressive disease after completion of radiotherapy.
  * No measurable lesion
  * Left ventricular ejection fraction (FEV) <50%
  * Diagnosis of any other malignancy during the last 5 years, except for in situ carcinoma of cervix uteri and squamous cell carcinoma of the skin
  * Any previous HER2 blocking therapy. Previous therapy with anti EGFR agents is allowed
  * Pregnancy or lactating
  * Other serious illness or medical condition including: Congestive heart failure (NYHA class II, III, IV) or history of documented congestive heart failure, unstable angina pectoris, myocardial infarction in the last 12 months, poorly controlled hypertension (systolic >180 mmHg or diastolic >100 mmHg), clinically significant valvular heart disease, or high-risk uncontrolled arrhythmias. Patients with dyspnoea at rest due to malignant or other disease (e.g. pulmonary metastases with lymphangitis) or who require supportive oxygen therapy. Active serious uncontrolled infections. Poorly controlled diabetes mellitus
  * Treatment with any investigational drug within 30 days before the beginning of treatment with study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Response rate | every two months

SECONDARY OUTCOMES:
Time to disease progression, overall survival, safety and assessment of biomarkers potentially implicated in trastuzumab sensitivity/resistance | every two months

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy